CLINICAL TRIAL: NCT06843421
Title: Korean Health Screening-Based Metabolic Dysfunction-Associated Steatotic Liver Disease Registry: A Retrospective Multicenter Cross-Sectional Study (K-MASLD Registry)
Brief Title: Korean Health Screening-Based Metabolic Dysfunction-Associated Steatotic Liver Disease Registry
Acronym: K-MASLD
Status: Not yet recruiting | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Hyung Joon Yim, Professor, Korea University
Other Study IDs: K-MASLD Registry
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Cardiovascular Diseases
Keywords: Metabolic Dysfunction-Associated Steatotic Liver Disease; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MASLD (Metabolic dysfunction-associated steatohepatitis) Group: Participants with fatty liver detected on abdominal ultrasound
- Normal Group: Participants with normal liver findings on abdominal ultrasound

SUMMARY:
The goal of this observational study is to establish a multi-center registry to better understand Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) using health screening data from Korean hospitals. MASLD is a liver condition where excess fat builds up in the liver and is closely linked to metabolic health problems like high blood pressure, diabetes, and obesity.

The main questions this study aims to answer are:

* What are the characteristics of people with MASLD?
* How is MASLD related to other health conditions, especially heart and blood vessel diseases?
* What factors might help identify MASLD early?

Researchers will compare two groups of people:

* People who have MASLD
* People who don't have MASLD (control group)

This study will look at health screening records from 2020 to 2023 from six Korean hospitals. The research team will collect and analyze:

* Basic health information (age, gender, weight, height, waist size)
* Lifestyle habits (drinking, smoking, exercise, eating habits)
* Medical conditions (high blood pressure, diabetes, high cholesterol)
* Results from medical tests including:

Liver ultrasound and Fibroscan results Heart CT scans Blood vessel ultrasound Blood test results Other health screening results

Participants in this study will not need to do anything new. The researchers will only look at information that was already collected during regular health screenings. All personal information will be protected and kept private.

This research could help doctors:

* Better understand who is at risk for MASLD
* Find MASLD earlier
* Develop better ways to prevent and treat MASLD
* Understand how MASLD is connected to other health problems

The study will take place over 3 years and includes adults age 19 and older who had health screenings at participating Korean hospitals. People who drink large amounts of alcohol or have other liver diseases will not be included in the study.

By learning more about MASLD through this registry study, researchers hope to improve healthcare for people with or at risk for this liver condition.

DETAILED DESCRIPTION:
Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is a condition characterized by excessive fat accumulation in the liver, associated with metabolic dysfunction. Unlike traditional concepts of Non-Alcoholic Fatty Liver Disease (NAFLD), MASLD emphasizes the central role of metabolic health in liver disease development. This condition is closely linked with metabolic syndrome components including insulin resistance, hyperglycemia, hypertension, and obesity. Patients with MASLD face increased risks of liver damage and functional decline, potentially progressing to liver fibrosis, cirrhosis, and even liver cancer. Additionally, MASLD shows strong associations with cardiovascular diseases, type 2 diabetes, and rheumatic conditions, making its management crucial for overall health maintenance.

The establishment of a multi-center registry for MASLD through Korean health screening data represents a significant advancement in liver disease research. The Korean healthcare system's comprehensive health screening infrastructure provides an exceptional opportunity to study MASLD systematically across multiple centers, as it routinely includes liver ultrasound, metabolic parameter assessments, and cardiovascular evaluations.

This study utilizes data from six major Korean hospitals to establish a detailed registry that will enhance our understanding of MASLD's characteristics and its associations with other health conditions. The liver's role as a central metabolic hub makes it crucial for studying the bidirectional relationship between hepatic function and systemic metabolic disorders. Recent evidence has shown strong connections between fatty liver disease and cardiovascular outcomes, making the inclusion of cardiac CT and carotid ultrasound data particularly valuable. Asian populations, including Koreans, often exhibit distinct patterns of MASLD compared to Western populations, particularly regarding body mass index thresholds and metabolic risk factors.

The registry implements innovative approaches to data collection and analysis by combining multiple data streams from routine health screenings, including advanced imaging techniques, metabolic parameters, inflammatory markers, cardiovascular risk factors, and lifestyle information. To ensure consistency across participating centers, the study employs standardized data collection protocols and unified formatting requirements, with centralized data management at Korea University Ansan Hospital.

The comprehensive approach to studying MASLD through health screening data represents a significant opportunity to advance our understanding of this condition in the Korean population. The findings from this registry will benefit current clinical practice and pave the way for future research and improvements in patient care. As metabolic health continues to be a growing concern globally, this registry's contributions to our understanding of MASLD will have far-reaching implications for public health and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* An individual who had an abdominal ultrasound performed

Exclusion Criteria:

* An individual with high alcohol intake history or other liver disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets adults aged 19 years and older who underwent health screenings at participating institutions from 2020 to 2023. The study population consists of subjects who had abdominal ultrasonography during their health screening, including those diagnosed with fatty liver (MASLD group, 500 subjects) and those with normal findings on ultrasonography (control group, 500 subjects) from each participating institution. Each of the 6 participating institutions will contribute 1,000 subjects (500 MASLD, 500 controls), for a total study population of 6,000 subjects. Subjects with high alcohol consumption or history of other liver diseases will be excluded from the study. All data will be collected and analyzed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Major Adverse Cardiovascular Events (MACE) | within 3 years
  MACE was defined as the composite endpoint of all-cause death, myocardial infarction, or stroke.

SECONDARY OUTCOMES:
Incidence Rate of Cancer | within 3 years
  Cancer was defined as the diagnosis of any malignant neoplasm during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung Joon Yim, MD., PhD., Principal Investigator — Korea University Ansan Hospital
Locations (5):
- South Korea (5):
  - Chung-Ang University Gwangmyeong Hospital, Gyeonggi-do, Gwangmyeong-si
  - Yonsei University Yongin Severance Hospital, Yongin, Gyeonggi-do
  - Inje Univerisity Sanggye Paik Hospital, Seoul, Nowon-gu
  - Wonju Severance Christian Hospital, Gangwon-do, Wonju-si
  - Ajou University Hospital, Suwon, Yeongtong-gu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong VW, Adams LA, de Ledinghen V, Wong GL, Sookoian S. Noninvasive biomarkers in NAFLD and NASH - current progress and future promise. Nat Rev Gastroenterol Hepatol. 2018 Aug;15(8):461-478. doi: 10.1038/s41575-018-0014-9. PMID 29844588
- [Background] Bedossa P, Patel K. Biopsy and Noninvasive Methods to Assess Progression of Nonalcoholic Fatty Liver Disease. Gastroenterology. 2016 Jun;150(8):1811-1822.e4. doi: 10.1053/j.gastro.2016.03.008. Epub 2016 Mar 19. PMID 27003601
- [Background] Angulo P, Kleiner DE, Dam-Larsen S, Adams LA, Bjornsson ES, Charatcharoenwitthaya P, Mills PR, Keach JC, Lafferty HD, Stahler A, Haflidadottir S, Bendtsen F. Liver Fibrosis, but No Other Histologic Features, Is Associated With Long-term Outcomes of Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2015 Aug;149(2):389-97.e10. doi: 10.1053/j.gastro.2015.04.043. Epub 2015 Apr 29. PMID 25935633
- [Background] Loomba R, Sanyal AJ. The global NAFLD epidemic. Nat Rev Gastroenterol Hepatol. 2013 Nov;10(11):686-90. doi: 10.1038/nrgastro.2013.171. Epub 2013 Sep 17. PMID 24042449
- [Background] Byrne CD, Targher G. NAFLD: a multisystem disease. J Hepatol. 2015 Apr;62(1 Suppl):S47-64. doi: 10.1016/j.jhep.2014.12.012. PMID 25920090
- [Background] Friedman SL, Neuschwander-Tetri BA, Rinella M, Sanyal AJ. Mechanisms of NAFLD development and therapeutic strategies. Nat Med. 2018 Jul;24(7):908-922. doi: 10.1038/s41591-018-0104-9. Epub 2018 Jul 2. PMID 29967350
- [Background] Tilg H, Moschen AR. Evolution of inflammation in nonalcoholic fatty liver disease: the multiple parallel hits hypothesis. Hepatology. 2010 Nov;52(5):1836-46. doi: 10.1002/hep.24001. PMID 21038418
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Rinella ME, Tacke F, Sanyal AJ, Anstee QM; participants of the AASLD/EASL Workshop. Report on the AASLD/EASL Joint Workshop on Clinical Trial Endpoints in NAFLD. Hepatology. 2019 Oct;70(4):1424-1436. doi: 10.1002/hep.30782. Epub 2019 Jul 9. PMID 31287572
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314